CLINICAL TRIAL: NCT07155187
Title: Phase 2/3 Open Label Randomized Study of Telisotuzumab Adizutecan Compared to Standard of Care in Subjects With Locally Advanced or Metastatic EGFR-Mutated Non-Squamous Non-Small Cell Lung Cancer After Progression on a Third-Generation EGFR TKI
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity of Intravenous (IV) Telisotuzumab Adizutecan Compared to Standard of Care in Adult Participants With Locally Advanced or Metastatic EGFR-Mutated Non-Squamous Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M25-713; 2025-521124-29 (Other: EU CT)
Record Dates: First submitted 2025-08-28; First posted 2025-09-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Telisotuzumab Adizutecan; ABBV-400, Standard of Care; Cancer; AndroMETa-Lung-713
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase 2: Telisotuzumab Adizutecan Dose A (Experimental): Participants will receive telisotuzumab adizutecan dose A, as part of the approximately 69 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan
- Phase 2: Telisotuzumab Adizutecan Dose B (Experimental): Participants will receive telisotuzumab adizutecan dose B, as part of the approximately 69 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan
- Phase 3: Telisotuzumab Adizutecan Recommended Phase 3 Dose (Experimental): Participants will receive telisotuzumab adizutecan at the recommended phase 3 dose, as part of the approximately 69 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan
- Phase 3: Stand of Care (SOC) (Experimental): Participants will receive investigator's choice of SOC, as part of the approximately 69 month study duration.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Telisotuzumab Adizutecan — Intravenous (IV) Infusion
  Arms: Phase 2: Telisotuzumab Adizutecan Dose A; Phase 2: Telisotuzumab Adizutecan Dose B; Phase 3: Telisotuzumab Adizutecan Recommended Phase 3 Dose
Drug: Standard of Care — Standard of Care
  Arms: Phase 3: Stand of Care (SOC)

SUMMARY:
Non-small cell lung cancer (NSCLC) is a common type of lung cancer where abnormal cells in the lungs grow out of control. The purpose of this study is to assess adverse events and change in disease activity of telisotuzumab adizutecan compared to standard of care (SOC).

Telisotuzumab adizutecan is an investigational drug being developed for the treatment of NSCLC. This study will be divided into two stages, in the first stage (phase 2) participants will receive 1 of 2 doses of telisotuzumab adizutecan. In the second stage (phase 3) participants will receive the recommended phase 3 dose (RP3D) of telisotuzumab adizutecan, from the previous stage, or SOC. Approximately 430 adult participants with NSCLC will be enrolled in the study in 200 sites around the world.

In phase 2, participants will receive 1 of 2 intravenous (IV) doses of telisotuzumab adizutecan. In phase 3, participants will receive the IV RP3D of telisotuzumab adizutecan, or SOC. The study will run for a duration of approximately 69 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of locally advanced or metastatic non-squamous non-small cell lung cancer (NSCLC) with documented EGFR Exon 19 deletion or Exon21 L858R mutation.
* Provide archived or recently obtained tumor tissue during Screening.
* Received one prior third-generation epidermal growth factor receptor tyrosine kinase inhibitor (EGFR TKI) therapy in the adjuvant, locally advanced, or metastatic setting, either as monotherapy or in combination with other agents, and experienced documented radiographic disease progression on or after therapy for the most recent regimen administered prior to study entry.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
* At least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, that has not been previously irradiated.
* Central nervous system (CNS) metastasis, these should be clinically asymptomatic or stable after definitive treatment.
* Current, historical, or suspected interstitial lung disease (ILD)/pneumonitis that required steroids should be excluded.
* If the prior third-generation EGFR TKI was administered in the adjuvant setting, progression must have occurred while on treatment.

Exclusion Criteria:

* Tumor(s) have adenosquamous or squamous histology or sarcomatoid features.
* Received more than 1 line of systemic therapy in the locally advanced or metastatic setting.
* Have any clinically significant medical conditions or any other reason that the investigator determines would interfere with the participant's participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Objective Response (OR) Assessed by Blinded Independent Central Review (BICR) | Up to Approximately 69 Months
  OR is defined as participants achieving a best overall response of confirmed complete response (CR) or confirmed partial response (PR) per BICR based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Phase 3: Progression-Free Survival (PFS) as assessed by BICR | Up to Approximately 69 Months
  PFS is defined as the time from randomization to the first occurrence of radiographic progression based on RECIST version 1.1 as determined by BICR or death from any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
Phase 2 and 3: Overall Survival (OS) as assessed by BICR | Up to Approximately 69 Months
  OS is defined as the time from randomization to the event of death from any cause.
Phase 2: PFS as assessed by BICR | Up to Approximately 69 Months
  PFS is defined as the time from randomization to the first occurrence of radiographic progression based on RECIST version 1.1 as determined by BICR or death from any cause, whichever occurs earlier.
Phase 2 and 3: Duration of Response (DoR) as Assessed by the BICR per RECIST v1.1 | Up to Approximately 69 Months
  DoR is defined as the time from the first response (CR or PR) to Progressive Disease (PD) or death (whichever occurs first) amongst confirmed responders.
Phase 2 and 3: Disease Control (DC) as Assessed by the BICR per RECIST v1.1 | Up to Approximately 69 Months
  DC is defined as best overall response of confirmed CR or confirmed PR, or stable disease (SD) based on RECIST, version 1.1.
Phase 3: OR Assessed by BICR | Up to Approximately 69 Months
  OR is defined as participants achieving a best overall response of confirmed CR or confirmed PR per BICR based on RECIST version 1.1.
Phase 3: Percentage of Participants with Change from Baseline in Physical Functioning as Measured by the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30) | Up to Week 12
  Health-related quality-of-life and symptoms will be assessed with the EORTC QLQ-C30, version 3.0. The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status (GHS)/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4 point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Phase 3: Percentage of Participants with Change from Baseline in Key Lung Cancer Symptoms as Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer Module 13 (EORTC QLQLC13) | Up to Week 12
  The EORTC QLQ-LC13 is a lung cancer specific module and consists of 13 questions assessing lung cancer-associated symptoms and treatment-related effects, including one multiple-item scale to assess dyspnea and a series of single items assessing coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain, and pain medication. Each item is assessed on a Likert scale from 1 (not at all) to 4 (very much).
Phase 3: Percentage of Participants with Change from Baseline in GHS/QoL as measured by the EORTC QLQ-C30 | Up to Week 12
  Health-related quality-of-life and symptoms will be assessed with the EORTC QLQ-C30, version 3.0. The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a GHS/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4 point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (23):
- United States (6):
  - Highlands Oncology Group - Springdale /ID# 277132, Springdale, Arkansas
  - Cancer Care Centers of Brevard- Rockledge /ID# 277853, Rockledge, Florida
  - Nho - Revive Research Institute /ID# 277569, Lincoln, Nebraska
  - Tennessee Cancer Specialists - Knoxville - Old Weisgarber Road /ID# 277891, Knoxville, Tennessee
  - SCRI Oncology Partners /ID# 276959, Nashville, Tennessee
  - Northwest Cancer Specialists - Vancouver /ID# 277855, Vancouver, Washington
- Australia (4):
  - Mater Hospital Brisbane /ID# 276985, South Brisbane, Queensland
  - Icon Cancer Centre Hobart /ID# 277549, Hobart, Tasmania
  - St Vincent's Hospital Melbourne /ID# 277002, Fitzroy, Victoria
  - Sunshine Hospital /ID# 276894, St Albans, Victoria
- Israel (5):
  - Meir Medical Center /ID# 277289, Kfar Saba, Central District
  - Rabin Medical Center /ID# 276748, Petah Tikva, Central District
  - Yitzhak Shamir Medical Center /ID# 276750, Ẕerifin, Central District
  - The Chaim Sheba Medical Center /ID# 276745, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus- Haifa /ID# 276746, Haifa
- Japan (4):
  - Hokkaido University Hospital /ID# 277240, Sapporo, Hokkaido
  - Kitasato University Hospital /ID# 277241, Sagamihara-shi, Kanagawa
  - National Cancer Center Hospital /ID# 277093, Chuo-Ku, Tokyo
  - Wakayama Medical University Hospital /ID# 277238, Wakayama, Wakayama
- South Korea (2):
  - Asan Medical Center /ID# 277371, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 277600, Seoul, Seoul Teugbyeolsi
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 277138, Kaohsiung City
  - Mackay Memorial Hospital /ID# 277146, Taipei

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-713